CLINICAL TRIAL: NCT05783271
Title: Validity of Parametric MRI Using VIRAD Scoring in the Diagnosis of Cancer Bladder
Brief Title: Validity of Parametric MRI Using VIRADS
Acronym: metricMRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, EmanTaha Abo-Elfadl, Validity of parametric MRI using VIRAD scoring in the diagnosis of cancer bladder, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: universty
Record Dates: First submitted 2023-03-02; First posted 2023-03-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mpMRI and biparametric MRI (Experimental): MRI images of the 58 patients with bladder tumors were transferred to a picture archiving communication system (PACS). The images were separated into two groups, namely set 1 (bp-MRI (non-contrast) protocol) and set 2 (mp-MRI protocol). Set 1 images has included three planes T2-WI and axial DWI sequences; set 2 images has included the DCE sequence in addition to set 1. Both of image sets were independently evaluated by a board-certified abdomi nal radiologist with 10 years of experience (reader 1) and general radiologist with 8 years of experience (reader 2). All lesions is scored in accordance with VI-RADS criteria in T2-WI, DWI, and DCE images separately, and the final VI-RADS score was determined. The lesions with VI-RADS scores 1-3 were evaluated as NMIBC, and VI-RADS scores 4 and 5 as MIBC .
  Interventions: Diagnostic Test: Gadolinium

INTERVENTIONS:
Diagnostic Test: Gadolinium — All patients will be subjected to :
  MRI examinations on a 1.5-T MRI system in the supine position by using a 16-channel pelvic phased-array coil. The MRI proto col includes the following sequences: unenhanced axial T1-WI, high-resolution three planes (axial, coronal, and sagittal) T2-WI, axial DWI with b values of 0, 800, and 1600 s/mm2, axial DCE T1-WI with three-dimensional (3D) high temporal resolution. In all sequences, the small field of view (FOV) was used with the scope of viewing the entire bladder, proximal urethra, distal ureteral orifices, and adjacent pelvic organs. Gadopentetate dimeglumine (Gadovist, 0.1 ml/kg body weight) is administered at a rate of 2 ml/s using a power injector.
  Other Names: MRI contrast

SUMMARY:
Our aim in this prospective study is to evaluate the validity of the non-contrast biparametric MRI (bp-MRI), including T2-WI and DWI sequences, and the availability of an alternative to the mp-MRI, for the muscle invasiveness assessment of bladder cancer using VIRAD scoring in both techniques.

DETAILED DESCRIPTION:
Urinary bladder cancer is the second most common neoplasm of the urinary tract worldwide. It accounts for 6-8% of malignancy in men and 2- 3% in women, with the highest incidence rates in North America , Europe and areas with endemic schistosomiasis in Africa and the Middle East.(1) Factors contribute to the development of bladder cancer are: advanced age, male sex, cigarette smoking and parasitic infection with schistosomiasis. Bladder cancer(BC)ranges from unaggressive non-invasive tumor(NMICB) that recur and commit patients to long life surveillance to aggressive and invasive tumors (MICB)with high disease mortality.(2) Knowledge of the clinical, histopathologic, and imaging features of common bladder neoplasms is essential.

The first-line imaging tool for assessing bladder lesions is ultrasonography, which may be followed by a computed tomography or magnetic resonance imaging if the origin of the mass is unclear or if distant spread is suspected.(3) Accurate preoperative diagnosis of detrusor muscle invasion of BC is important because non- muscle-invasive (stage T1 or lower) and muscle-invasive (stage T2 or higher) BC are treated differently.Prognosis of the tumor depends mainly on grade ,depths of invasion and the presence of carcinoma insitu(CIS).(4) MRI now become the modality of choice for the local staging of BC , assessment of regional lymph node involvement and the tumor spread to pelvic bones and upper urinary tract.(5) As it has high tissue contrast, multiplanar imaging capabilities, and the ability of tissue characterization.(6) Currently, the multi-parametric magnetic resonance imaging (mp-MRI) is widely used for bladder cancer diagnosis and staging. It consists of the conventional sequence [T2-weighted anatomic imaging (T2WI)] and functional MRI techniques [dynamic contrast-enhanced (DCE) imaging and diffusion-weighted imaging (DWI)] .(7).With diagnostic accuracy in differentiation between MICB and NMICB was 84% with highest sensitivity 78%.(9) DWI used in mp-MRI is reported as the dominant sequence in evaluating BC muscle invasion .(14) To Avoid contrast material-related complications,the question askesd : Is contrast material important in the local staging of BC ?( 13) So assessing the diagnostic validity of the non contrast biparametric MRI (bpMRI) with that of (mpMRI) based on the Vesicle Imaging-Reporting and Data System (VI-RADS) in predicting muscle invasion by bladder cancer (BCa) is needed.(10). (VIRADS) scoring system was created in 2018 to standardise imaging and reporting of bladder cancer staging with mp- MRI which suggests the likelihood of detruser muscle invasion. Muscle invasion disease carries a worse prognosis and requires radical surgery.(4) VI-RADS provides high diagnostic accuracy to diagnose high grade and muscle invasive bladder cancer.(11)

:Prospectively calculated and collected data will be analysed. Computer software: SPSS package 23 Statistical tests: Descriptive statistics will be performed with frequency and cross tabulations for categorical variables. Means and standard deviations will be measured for numerical variables. The chi-square test will be used for comparing independent categorical variables. Monte Carlo simulations will be run for multiple groups if comparisons will not meet the chi-square criteria; Fishers exact test will be used in the comparison of the groups. Students t-test will be used for comparing the numerical data displaying normal distribution; the MannWhitney U-test will be performed for the numerical variables not displaying normal distribution. The P-value will be set at 0.05 and all of the comparisons will be two-tailed.

ELIGIBILITY:
Inclusion Criteria:

58 cases of patients who suspected to have cancer urinary bladder by clinical, histopathological examination and radiological imaging.

All age groups . Both sex

Exclusion Criteria:

patient with high renal chemistry. Patient with contraindications to MRI as pacemaker and cochlear implants.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess validity of parametric MRI in terms of accuracy and validity using VIRAD scoring in the diagnosis of cancer bladder | 2 years
  in this cohort study ,we will examine patients refered to radiology department Assuit university hospital by mpMRI from 1/3/2025 untill 31/12/2026 then all data will be regrouped to know: Is bi-parametric-MRI protocol has a diagnostic accuracy comparable to an mp-MRI protocol for the detection of muscle invasive BC using the VI-RADS criteria.
Validity | 2 years
  Aiming for high specificity or sensitivity to achieve the best patient results

CONTACTS AND LOCATIONS:
Overall Officials: Hassan A.Abolella, Proff, Principal Investigator — Newvalley University
Locations (1):
- Assuit university, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saginala K, Barsouk A, Aluru JS, Rawla P, Padala SA, Barsouk A. Epidemiology of Bladder Cancer. Med Sci (Basel). 2020 Mar 13;8(1):15. doi: 10.3390/medsci8010015. PMID 32183076
- [Background] Lenis AT, Lec PM, Chamie K, Mshs MD. Bladder Cancer: A Review. JAMA. 2020 Nov 17;324(19):1980-1991. doi: 10.1001/jama.2020.17598. PMID 33201207
- [Background] Shelmerdine SC, Lorenzo AJ, Gupta AA, Chavhan GB. Pearls and Pitfalls in Diagnosing Pediatric Urinary Bladder Masses. Radiographics. 2017 Oct;37(6):1872-1891. doi: 10.1148/rg.2017170031. PMID 29019749
- [Background] Wang H, Luo C, Zhang F, Guan J, Li S, Yao H, Chen J, Luo J, Chen L, Guo Y. Multiparametric MRI for Bladder Cancer: Validation of VI-RADS for the Detection of Detrusor Muscle Invasion. Radiology. 2019 Jun;291(3):668-674. doi: 10.1148/radiol.2019182506. Epub 2019 Apr 23. PMID 31012814
- [Background] Rabie E, Faeghi F, Izadpanahi MH, Dayani MA. Role of Dynamic Contrast-Enhanced Magnetic Resonance Imaging in Staging of Bladder Cancer. J Clin Diagn Res. 2016 Apr;10(4):TC01-5. doi: 10.7860/JCDR/2016/17596.7690. Epub 2016 Apr 1. PMID 27190913
- [Background] Caglic I, Panebianco V, Vargas HA, Bura V, Woo S, Pecoraro M, Cipollari S, Sala E, Barrett T. MRI of Bladder Cancer: Local and Nodal Staging. J Magn Reson Imaging. 2020 Sep;52(3):649-667. doi: 10.1002/jmri.27090. Epub 2020 Feb 29. PMID 32112505
- [Background] Panebianco V, Narumi Y, Altun E, Bochner BH, Efstathiou JA, Hafeez S, Huddart R, Kennish S, Lerner S, Montironi R, Muglia VF, Salomon G, Thomas S, Vargas HA, Witjes JA, Takeuchi M, Barentsz J, Catto JWF. Multiparametric Magnetic Resonance Imaging for Bladder Cancer: Development of VI-RADS (Vesical Imaging-Reporting And Data System). Eur Urol. 2018 Sep;74(3):294-306. doi: 10.1016/j.eururo.2018.04.029. Epub 2018 May 10. PMID 29755006
- [Background] Del Giudice F, Flammia RS, Pecoraro M, Moschini M, D'Andrea D, Messina E, Pisciotti LM, De Berardinis E, Sciarra A, Panebianco V. The accuracy of Vesical Imaging-Reporting and Data System (VI-RADS): an updated comprehensive multi-institutional, multi-readers systematic review and meta-analysis from diagnostic evidence into future clinical recommendations. World J Urol. 2022 Jul;40(7):1617-1628. doi: 10.1007/s00345-022-03969-6. Epub 2022 Mar 16. PMID 35294583
- [Background] Makboul M, Farghaly S, Abdelkawi IF. Multiparametric MRI in differentiation between muscle invasive and non-muscle invasive urinary bladder cancer with vesical imaging reporting and data system (VI-RADS) application. Br J Radiol. 2019 Dec;92(1104):20190401. doi: 10.1259/bjr.20190401. Epub 2019 Oct 8. PMID 31573328
- [Background] Noh TI, Shim JS, Kang SG, Sung DJ, Cheon J, Sim KC, Kang SH. Comparison between biparametric and multiparametric MRI in predicting muscle invasion by bladder cancer based on the VI-RADS. Sci Rep. 2022 Nov 30;12(1):20689. doi: 10.1038/s41598-022-19273-7. PMID 36450813
- [Background] Gmeiner J, Garstka N, Helbich TH, Shariat SF, Baltzer PA. Vesical Imaging Reporting and Data System (VI-RADS): Are the individual MRI sequences equivalent in diagnostic performance of high grade NMIBC and MIBC? Eur J Radiol. 2021 Sep;142:109829. doi: 10.1016/j.ejrad.2021.109829. Epub 2021 Jun 24. PMID 34252867
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Delli Pizzi A, Mastrodicasa D, Taraschi A, Civitareale N, Mincuzzi E, Censi S, Marchioni M, Primiceri G, Castellan P, Castellucci R, Cocco G, Chiacchiaretta P, Colasante A, Corvino A, Schips L, Caulo M. Conspicuity and muscle-invasiveness assessment for bladder cancer using VI-RADS: a multi-reader, contrast-free MRI study to determine optimal b-values for diffusion-weighted imaging. Abdom Radiol (NY). 2022 May;47(5):1862-1872. doi: 10.1007/s00261-022-03490-9. Epub 2022 Mar 18. PMID 35303112
- [Background] Aslan S, Cakir IM, Oguz U, Bekci T, Demirelli E. Comparison of the diagnostic accuracy and validity of biparametric MRI and multiparametric MRI-based VI-RADS scoring in bladder cancer; is contrast material really necessary in detecting muscle invasion? Abdom Radiol (NY). 2022 Feb;47(2):771-780. doi: 10.1007/s00261-021-03383-3. Epub 2021 Dec 17. PMID 34919161